CLINICAL TRIAL: NCT00002433
Title: Activation of Alveolar Macrophages by Aerosolized r-metHuIFN-Gamma (IFN-Gamma) in Patients With AIDS
Brief Title: The Effects of r-metHuIFN-Gamma on the Lungs of Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amgen (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 062A; IFNG-8901
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-11

CONDITIONS: HIV Infections
Keywords: Pulmonary Alveoli; Macrophage Activation; Interferon-gamma, Recombinant; Injections, Subcutaneous; Aerosols; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — interferon gamma-1b

INTERVENTIONS:
Drug: Interferon gamma-1b

SUMMARY:
To determine safety and tolerance of administering aerosolized recombinant interferon gamma (IFN-gamma) for 4 weeks in patients with AIDS. To examine activation of alveolar macrophages by aerosolized IFN-gamma administration. To determine if subcutaneous (SC) injection of IFN-gamma can activate alveolar macrophages in AIDS patients.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Diagnosis of AIDS with one or more opportunistic infections.
* Kaposi's sarcoma with prior history of opportunistic infection.
* Stable dose of zidovudine (AZT) therapy.
* Preserved pulmonary, renal and hepatic function.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Presence of active infection.
* Active opportunistic infections.
* Cardiac disease.
* Central nervous system disorders.
* History of seizures.
* Irreversible airway disease.

Patients with the following are excluded:

* Co-existing conditions and symptoms listed in Patient Exclusion Co-existing Conditions.

Prior Medication:

Excluded within 4 weeks of study entry:

* Immunosuppressive therapy.
* Cytotoxic therapy.
* Excluded:
* Interferon gamma therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Locations (1):
- New York Hosp - Cornell Med Ctr, New York, New York, United States